CLINICAL TRIAL: NCT05252325
Title: Prospective, Controlled, Randomized, Blinded Evaluator, Split-face Clinical Study to Evaluate the Efficacy and Safety of Hyaluronic Acid Hydrogel With Lidocaine Lidocaine for the Treatment of Moderate to Severe Nasolabial Folds
Brief Title: Clinical Study on Hyaluronic Acid With Lidocaine for the Treatment of Moderate to Severe Nasolabial Folds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centro Medico Polispecialistico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HA28L/MD01/20
Record Dates: First submitted 2022-01-20; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Nasolabial Folds

STUDY DESIGN:
Intervention Model Description: pre-CE mark controlled, prospective, randomized, blinded evaluator, single centre, split-face clinical investigation
Who Masked: Outcomes Assessor
Masking Description: The products will be administered by the Investigator/Co-Investigator (Treating Investigator), while the evaluations will be done by a Co-Investigator not aware of the side type treatment (Blinded Evaluator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAL on the right side of the face; HA on the left side of the face (Other): the subjects will receive HAL ( hyaluronic acid +lidocaine)in the right side of the face, HA (hyaluronic acid without lidocaine) in the left side
  Interventions: Device: hyaluronic acid plus lidocaine; Device: hyaluronic acid without lidocaine
- HAL on the left side of the face; HA on the right side (Other): the subjects will receive HA in the right side of the face, HAL in the left side
  Interventions: Device: hyaluronic acid plus lidocaine; Device: hyaluronic acid without lidocaine

INTERVENTIONS:
Device: hyaluronic acid plus lidocaine — local injection for correction of nasolabials fold
Device: hyaluronic acid without lidocaine — local injection for correction of nasolabial folds

SUMMARY:
This will be a pre-CE mark controlled, prospective, randomized, blinded evaluator, single centre, split-face clinical investigation.

Each subject will receive both medical devices under investigation, one (HAL: Hyaluronic Acid plus Lidocaine ) on the one side of the face, the other (HA: Hyaluronic Acid) on the other side, in randomized fashion.

DETAILED DESCRIPTION:
This will be a pre-CE mark controlled, prospective, randomized, blinded evaluator, single centre, split-face clinical investigation.

Each subject will receive both medical devices under investigation, one (HAL) on the one side of the face, the other (HA) on the other side, in randomized fashion.

The products will be administered by the Investigator/Co-Investigator (Treating Investigator), while the evaluations will be done by a Co-Investigator not aware of the side type treatment (Blinded Evaluator).

The investigational plan include a Visit 1, during which subjects will be screened for entry (inclusion/exclusion) criteria; eligible subjects will be treated with the medical devices and followed for the next hour for pain and safety evaluation.

Visit 2, 3 and Visit 4 are schedule after 2 (± 2 days), 12 (± 10 days) e 24 (± 10 days) weeks for the assessment of safety and clinical efficacy.

Subjects prematurely discontinued from the investigation after the treatment will perform an 'Early termination visit', in which procedures scheduled for Visit 4 (24 weeks, final visit) will be performed (whenever feasible). In case of premature discontinuation of the investigation, the Investigator will duly record the reason for premature withdrawal in the appropriate section of the case report form (CRF).

Visit 4 (or the 'Early termination Visit') will represent the conclusion of subject's participation in the investigation.

Adverse events will be recorded during the entire investigational period by investigator's assessment and subjects' spontaneous reporting. Vital signs (blood pressure and heart rate) will be measured at each visit in the investigational site

ELIGIBILITY:
Inclusion Criteria:

* Presence of moderate to severe nasolabials folds (WSRS grade 3-4);
* Reasonable potential benefit from correction;
* Subjects able to understand the full nature and the purpose of the investigation, including possible risks and side effects, able to cooperate with the Investigator and to comply with the requirements of the entire investigation (ability to attend all the planned investigation visits according to the time limits included) based on Investigator's judgement;
* Subjects must voluntarily give written informed consent, adhere to the protocol and report events and concomitant medication for the entire duration of investigation.

Exclusion Criteria:

* Pregnant (as determined by a urine pregnancy test at the screening visit) or lactating women. For the entire duration of the investigation, female subjects of childbearing potential (i.e., not permanently sterilised - post hysterectomy or tubal ligation status - or not postmenopausal from at least one year) must adopt an appropriate method of contraception according to the definition of Note 3 of ICH M3 Guideline;
* Prior treatment of the face (e.g. other permanent or biodegradable injectable fillers or surgical correction such as a face-lift, etc.) within 3 months prior to entry into the study or planned to undergo such therapy during the study;
* Previous tissue augmentation with permanent implants (e.g., silicone) in the area to be treated;
* Presence of active inflammation, infection (acne, herpes, dermatitis, etc.) or unhealed wound of the face;
* Presence of varices in the area to be treated;
* History of hypertrophic scarring;
* Medical history or clinical examination positive for metabolic or endocrine serious diseases (e.g. uncontrolled diabetes or diabetes complications), anaphylaxis, severe allergies, immune disorders affecting the skin, other local or systemic concomitant diseases that may interfere with healing or with protocol evaluation parameters;
* Use of non-steroidal anti-inflammatory drugs (NSAIDs), analgesics, antiplatelets and anticoagulants in the week before treatment;
* Use of any other treatment or medication that, according to its pharmacological properties and in the opinion of the Investigator, can alter the perception of pain, started in the week before the screening visit;
* Use of narcotic agents, antineoplastics, immunosuppressants or of any other agent that may interfere with healing in the 4 weeks before the screening visit;
* Neurological or psychiatric diseases that may threaten the obtaining of informed consent or the adherence to investigation procedures;
* Ongoing neoplastic (including skin cancer) and/or immunodepressive diseases;
* Subjects with known allergy or hypersensitivity to at least one component of any of the investigational medical devices;
* Ongoing or scheduled during the study radiation, laser, ultrasound, chemical peels treatment in the target area;
* Known hypocoagulability state;
* History of drugs and/or alcohol abuse;
* Subjects unable to measure pain properly by means of a visual analogue scale (VAS);
* Subjects considered to be unsuitable to participate, in the investigators opinion, for any other reason;
* Planned relocation during the study, which would make follow-up visits impossible;
* Concomitant participation in other clinical investigations or participation in the evaluation of any investigational drugs/devices during 3 months before this investigation or previous participation in the same investigation or planned to receive other investigational products during the study .

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
changes in pain due to the injection assessed by VAS (Visual Analogue Scale, 0-100 mm) at 15-30-45-60 minutes after each injection(baseline) | within 1 min and 15-30-45-60 minutes after each injection
  pain experienced by subjects during and immediately after injections of the products under investigation [hyaluronic acid PEG-cross-linked formulated with 0.3% lidocaine: HAL] versus the same product WITHOUT lidocaine [HA], separately for each side of the face. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Clinical efficacy | done by the subject at weeks 2, 12 and 24 after treatments, separately for each side of the face
  Global Aesthetic Improvement Scale (GAIS):
  very much improved: excellent corrective result; much improved: marked improvement of the appearance, but not optimal; improved: improvement of the appearance, better compared with the initial condition, but a touch-up is advised; no change: the appearance substantially remains unchanged in respect of the original condition; worse: the appearance worsened compared with the initial condition.
Clinical efficacy | done by the blind evaluator before intervention and 12-24 weeks after injections, separately for each side of the face
  Wrinkle Severity Rating Scale (WSRS):
  1. absent- no visible nasolabial fold; continuous skin line
  2. mild - shallow but visible nasolabial fold with a slight indentation; minor facial feature; implant is expected to produce a slight improvement in appearance
  3. moderate- moderately deep nasolabial fold; clear facial feature visible at normal appearance but not when stretched; excellent correction is expected from injectable implant
  4. severe- very long and deep nasolabial fold; prominent facial feature; <2 mm visible fold when stretched; significant improvement is expected from injectable implant
  5. extreme- extremely deep and long nasolabial fold, detrimental to facial appearance; 2-4 mm visible V-shaped fold when stretched; unlikely to have satisfactory correction with injectable implant alone
Clinical efficacy | done by the blind evaluator and by the the subject at the week 24 of the study, separately for each side of the face
  Global satisfaction assessment (GSA) scale:
  unsatisfying satisfying very satisfying

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/25/NCT05252325/Prot_SAP_000.pdf